CLINICAL TRIAL: NCT03187171
Title: Comparison of Outcomes After ACDF Using Allograft Fusion Versus PEEK Fusion: a Prospective Clinical Trial
Brief Title: ACDF Comparison Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083342
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Cervical Spine Disc Disease; Surgery; Fusion of Spine; Degenerative Disc Disease
Keywords: Anterior Cervical Spine Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized comparative outcomes study, in which all subjects who fit the inclusion and exclusion criteria and who agreed to be part of the study will be randomized to either Allograft or Cohere PEEK fusion group and will be followed for approximately 12 months following surgery according to the standard-of-care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Allograft Fusion Group (Active Comparator): The anterior approach to the cervical spine for discectomy and fusion by the insertion of an autologous iliac crest tricortical bone graft.
  Interventions: Other: Allograft Fusion
- Cohere PEEK Fusion Group (Active Comparator): The anterior approach to the cervical spine for discectomy and fusion by the insertion of a Cohere porous PEEK fusion device.
  Interventions: Device: Cohere PEEK Fusion Group

INTERVENTIONS:
Other: Allograft Fusion — ACDF is a surgical technique used to treat a variety of cervical spine disorders, such as nerve root or spinal cord compression, cervical spondylosis, and cervical spinal stenosis. The anterior approach to the cervical spine for discectomy and fusion by the insertion of an autologous iliac crest tricortical bone graft was first described by Robinson and Smith in 1955. In 1958, Cloward described a wide anterior cylindrical discectomy performed with a special reamer combined with anterior fusion by the insertion of autologous iliac bone graft of the same shape. At Duke University Health Systems, both allografts and Cohere porous PEEK fusion device are used for ACDF.
  Arms: Allograft Fusion Group
Device: Cohere PEEK Fusion Group — Bagby et al. developed the first interbody fusion cage. Cages of different shapes and materials are used to perform ACDF which, in some cases, could be associated with plate fixation. At Duke University Health Systems, both allografts and Cohere porous PEEK fusion device are used for ACDF.
  Other Names: Fusion Device; PEEK Cage
  Arms: Cohere PEEK Fusion Group

SUMMARY:
This research protocol seeks to compare radiological and clinical outcomes of cervical spine disease patients following standard-of-care anterior cervical discectomy and fusion (ACDF) using allograft fusion versus Cohere porous polyetheretherketone (PEEK) fusion device.

This clinical study presents little to no additional risk to study subjects beyond those associated with standard-of-care ACDF surgery. Adults age 18 and over who are undergoing an ACDF procedure will be enrolled in the study. The study consists of a completing a series of questionnaires and obtaining radiographs. The primary endpoint of the study will be the rate of successful spinal fusion for each group. For evaluation of the primary endpoint and additional assessments, descriptive statistics including mean, standard deviation, minimum, median, and maximum for continuous variables and frequency distribution for categorical variables will be provided, as well as tabular listings. All complications will be itemized including incidence, duration, and relationship to the device used and/or procedures performed.

DETAILED DESCRIPTION:
This is a prospective randomized comparative outcomes study, in which all subjects who fit the inclusion and exclusion criteria and who agreed to be part of the study will be randomized to either Allograft or Cohere polyetheretherketone (PEEK) fusion group and will be followed for approximately 12 months following surgery according to the standard-of-care.

Pain and function will be assessed using neck disability index (NDI), 36-Item Short Form Survey (SF-36), and Numeric Rating Scale (NRS). A trained study team member will record a standardized neurologic examination, including motor, sensory, and reflexes. Neurologic success is defined as maintenance or improvement of all 3 neurologic parameters (motor, sensory, and reflexes). The clinical results will also be assessed using the Japanese Orthopedic Association (JOA) scoring system for cervical myelopathy.

Flexion and extension radiographs will be obtained pre-operatively, at 6-months and 12-months after surgery. A CT scan will be obtained at 6 months, if fusion has occurred no CT is needed at 12 months, if fusion did not occur another computerized tomography (CT) scan will obtained at 12 months. From previous literature, successful fusion is defined as ≤2° of angular motion on lateral flexion and extension radiographs, the presence of bridging trabecular bone between the vertebrae being fused, and the absence of any radiolucent zones spanning more than 50% of the allograft surface. Two independent blinded radiologists will assess the radiographs. In the event of disagreement about fusion healing, a third independent reading will be obtained from a third radiologist.

ELIGIBILITY:
Inclusion Criteria:

1. 18 or more years of age
2. Able to provide informed consent
3. Has documented diagnosis of cervical spine radiculopathy and/or myelopathy
4. Is undergoing standard-of-care ACDF

Exclusion Criteria:

1. Prior cervical spine surgery
2. Single-level ACDF
3. Has a systemic infection or cervical spine infection
4. Has a medical condition that may interfere with bone and soft tissue healing
5. Any condition that, in the opinion of the investigator, may preclude accurate data collection or evaluation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Rate of successful fusion. | 18 months
  To compare post-operative bone fusion following standard-of-care ACDF using allograft fusion or Cohere porous PEEK fusion.

SECONDARY OUTCOMES:
Overall success rate - composite score. | 18 months
  To be considered an overall success, patients have to achieve all of the following: a ≥15 point improvement in their NDI scores, maintenance or improvement in their neurologic status, no serious adverse events related to the implant or surgical procedure, and no subsequent surgery or intervention that is classified as "failure."

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haglund, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No